CLINICAL TRIAL: NCT05632510
Title: PREVENTION OF PERINATAL DEPRESSION BY EPDS DURING THE FIRST PRENATAL CONSULTATION AT MATERNITY DEPARTMENT: A CLUSTER-RANDOMIZED CONTROLLED TRIAL
Brief Title: PREVENTION OF PERINATAL DEPRESSION BY EPDS DURING THE FIRST PRENATAL CONSULTATION AT MATERNITY DEPARTMENT
Acronym: PREVIDEPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: APHP200025; 2020-A03097-32 (Other: ID-RCB)
Record Dates: First submitted 2022-10-31; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-10

CONDITIONS: Peripartum Depression (PPD)

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPDS Group (Other)
  Interventions: Diagnostic Test: The Edinburgh Postnatal Depression Scale (EPDS)
- Courent practice Group (No Intervention)

INTERVENTIONS:
Diagnostic Test: The Edinburgh Postnatal Depression Scale (EPDS) — The Edinburgh Postnatal Depression Scale (EPDS) is a self-administered questionnaire of 10 items, is recommended by the NICE guideline and French National Authority for Health for screening peripartum women, validated in French and well accepted.
  Arms: EPDS Group

SUMMARY:
The risk of PPD for a woman giving birth ranges between 10 and 20% worldwide, with about a third of postpartum depression that begin during pregnancy. PPD has been associated to negative short-/long-term effects for the mother's health, the child's health and early interactions when left untreated.

PPD is underdiagnosed, less than half of patients being diagnosed partly because of atypical symptoms, reluctance of patients to seek help, and because of the lack of systematic screening for this condition. Other specific biological changes could also be involved. Reduction in plasma oxytocin levels have been shown to be associated with the risk of PPD and heritability studies have identified a genetic contribution.

The Edinburgh Postnatal Depression Scale (EPDS) is a self-administered questionnaire of 10 items, is recommended by the NICE guideline and French National Authority for Health for screening peripartum women, validated in French and well accepted.

In France, the first contact with midwives or obstetricians during pregnancy usually occurs around the 4th month of pregnancy. French National Authority for Health recommends evaluation of risk factors for depression during this first consultation. However, this interview is rarely done probably because assessment of depression could be considered as difficult and time consuming. However, a meta-analysis shows that screening depression in the general population significantly reduces the risk for persistent depression (relative risk 0.87 [95%CI 0.79 to 0.95]), as compared to usual care.

Our hypothesis is that early identification of vulnerability/depression in pregnant women would enable clinical team to offer adequate psychological and psychosocial care during pregnancy, thus reducing PPD in these women.

The investigators propose to assess the impact of a systematic screening of depression using EPDS during an early consultation in comparison with usual practices, on the risk of depression during peripartum period (PPD).

DETAILED DESCRIPTION:
Follow-up of pregnancy by medical staff will be performed as usual: referral to specific structures, according to the usual hospital care protocols, which do not fall within the scope of this protocol.

An independent psychologist will conduct blinded evaluation of perinatal depression using a semi-structured interview (DIGS) based on the DSM-5 criteria (i) between the first and fifth day postpartum and (ii) at 8 weeks post-partum to assess the primary endpoint. The interview will also allow assessment of management of specialized care during pregnancy and during postpartum at week 8 after childbirth (specialized consultation, psychotherapy, drug treatment: nature, frequency and doses for therapeutics).

The choice of a cluster randomization over individual randomization is justified by the risk of contamination bias in the depression screening. The choice of a clinician randomization over center randomization is justified by the high heterogeneity of patient's characteristics between centres.

ELIGIBILITY:
Inclusion Criteria:

Adult women (aged > 18 years)

* Between 10 and 24 weeks pregnancy
* Fluent in written and spoken French (can understand a self-administered questionnaire);
* Affiliated to a social security scheme
* Informed consent obtained

Exclusion Criteria:

* Reported diagnosis of schizophrenia or physical and intellectual state incompatible with a clinical evaluation
* Persons unable to give their consent
* Unable adults (maintenance of justice, tutelage, legal guardianship)
* Person deprived of her liberty
* Patient on AME (state medical aid)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 4471 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
The perinatal major depressive episode during the period starting at 8 weeks before childbirth and ending 8 weeks postpartum. | 8 weeks before childbirth and 8 weeks postpartum
  To show the superiority of the implementation of the Edinburgh Postnatal Depression Scale (EPDS) as a depression screening tool during early pregnancy consultation, compared with usual depression screening to reduce the risk of peripartum depression.
  The primary endpoint is the diagnosis of a depressive episode according to DSM-5 criteria during the period from 8 weeks before childbirth to 8 weeks postpartum.

SECONDARY OUTCOMES:
Antenatal (from 8 weeks before delivery to delivery) major depressive episode as defined by the DSM-5 criteria | 8 weeks before childbirth and 8 weeks postpartum
  assessed between the first and fifth days after birth.by a face-to-face interview conducted by a psychologist, using the DIGS
Prevalence of a postpartum (from delivery to 8 weeks postpartum) major depressive episode as defined by the DSM-5 criteria | childbirth and 8 weeks postpartum
  assessed at 8 weeks postpartum by a phone interview, conducted by a psychologist, using the DIGS
Specific care received by women from childbirth to 8 weeks after delivery | childbirth and 8 weeks postpartum
  It will be assessed at the maternity department, by a face-to-face interview conducted by a psychologist.
Specific care received by women from childbirth to 8 weeks after delivery | childbirth and 8 weeks postpartum
  (specialized consultation, psychotherapy, drug treatment, hospitalization in psychiatry, etc : nature, frequency, doses if therapeutics). It will be assessed by a phone interview, conducted by a psychologist.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline DUBERTRET, Principal Investigator — Assistance Publique - Hôpitaux de Paris (AP-HP)
Locations (1):
- Louis Mourier hospital, Colombes, France